CLINICAL TRIAL: NCT06630533
Title: Effect of Baduanjin on Balance and Fall Risk in Elderly Individuals
Brief Title: Effect of Baduanjin in Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, alyildirim, Principal Investigator, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 145353
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Exercise
Keywords: exercise; functional balance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin Exercise Group (Experimental): The experimental group received Baduanjin training for 8 weeks (5 days a week). Baduanjin training was given face-to-face 3 days a week by a physiotherapist who is a Baduanjin trainer. Participants practiced it at home as a home exercise 2 days a week.
  Interventions: Other: Baduanjin Exercise Group
- Control Group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Baduanjin Exercise Group — Baduanjin exercises (Eight-Part Exercises or Eight-Part Brocades), an important part of Qigong, consist of eight postures (1-holding the hands high with palms up, 2- posing as an archer shooting, 3- holding one arm aloft, 4- looking backwards, 5- swinging the head and lowering the body, 6- moving the hands down the back and legs and touching the feet, 7- thrusting the fists and making the eyes glare, and 8- raising and lowering the heels).
  Arms: Baduanjin Exercise Group

SUMMARY:
Aging is a biological process that begins with the birth of individuals and continues until death. With increasing age, the human body enters a process in which structural and functional changes occur and may differ between individuals. This study aims to determine the effect of Baduanji by reducing or completely eliminating the risk of loss of balance and falls in elderly individuals. 60 people between the ages of 65-85 will be included in the study. Individuals will be randomly divided into two groups. In the study, the Berg Balance Scale (BDS) was used to assess balance and the Timed Up and Go Test (TUGT) test was used to assess functional levels. In our study, the Baduanjin exercise program will be applied 5 days a week for 8 weeks with the supervision of a physiotherapist. The Baduanjin exercise program will be applied to the first group, the second group will be the control group and no intervention will be made.

DETAILED DESCRIPTION:
Aging is a biological process that begins with the birth of individuals and continues until death. With advancing age, the human body enters a process in which structural and functional changes occur and may differ between individuals. Approximately 50-75% of individuals over the age of 65 experience balance and ambulation problems. Balance in living things is the ability to keep the body gravity line within stability limits and to maintain this. Balance disorders can be seen as a result of pathological disorders such as neurological diseases, sensory disorders or muscle weakness, as well as the loss of muscle strength and sensory functions observed during the normal aging process or the decrease in the speed of sensory motor responses. Although the balance system in humans is at an optimal level in early adulthood, deteriorations are observed after approximately the age of 50. In recent years, the importance of physical activity has begun to be emphasized more in order to remind individuals that they are a productive part of society in old age, to minimize the inadequacies, disabilities and discomforts that occur with aging, and to enable them to continue their lives independently. Physical activity is central to most programs designed to reduce the risk of falling and can work with strength, balance, and other physiological and psychological pathways. When the literature is examined, current studies have shown that older individuals have positive perspectives on traditional aerobic exercise. Tai Chi has been proven to improve balance and physical function. Qigong, which emerged before Tai Chi, is considered another traditional aerobic exercise preferred by older individuals who are intolerant of intense physical activities. Baduanjin exercise (Eight-Part Exercises or Eight-Part Brocades), an important complementary part of Qigong, consists of eight separate postures (supporting the chest, drawing bows to both sides, lifting one hand, practicing looking back, waving the hand and wagging the tail, touching the feet with both hands, climbing with both hands, and relaxing your back). Baduanjin is a series of exercises that are a qigong (chi kung) practice of Chinese origin. The term "Ba Duan Jin" means "eight pieces of brocade" or "eight silk ropes" in Chinese. This exercise series includes a series of movements that include body posture, breath control, and mental concentration. The main purpose of Baduanjin is to increase energy (chi or qi) circulation, provide balance in the body, increase flexibility, and improve overall health. According to traditional Chinese medicine, the free circulation of chi and its balanced distribution in the body are the keys to a healthy life. This exercise series aims to create a balance in physical, mental, and energetic terms. Each of them can have beneficial effects on different parts of the body or specific organs. Similar to Tai Chi, Baduanjin exercise is also considered a multi-component therapy that combines physical, psychosocial, cognitive, and spiritual components. Compared to Tai Chi, Baduanjin exercise has fewer physical and cognitive requirements, making it very suitable for short-term application in elderly individuals. In this context, the study aims to determine the effect of Baduanjin by reducing or completely eliminating the risk of loss of balance and falls in elderly individuals, and aims to shed light on future studies.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 65-85,
* being a volunteer to participate in the study, -having a good enough cognitive level to understand the questions in the evaluation form, --
* being able to stand independently.

Exclusion Criteria:

* having any musculoskeletal system problem that would affect walking and balance,
* having a hearing problem that could impair communication,
* having severe visual problems,
* having a history of injury in the last 6 months,
* having undergone lower extremity surgery such as hip-knee replacement.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 8 weeks
  The Timed Up & Go (TUG) Test : The timed up and go test was used for functional assessment of the patients. This test is important in terms of testing the patients' ability to maintain balance as well as evaluating their walking speed.
Primary Outcome Measure: | 8 weeks
  Berg balance test is a scale developed to measure the balance of elderly individuals. With the Berg balance test, 14 functions are evaluated throughout the test and the scores given to the patient are added up at the end of the test. As a result, the evaluated person receives a score between 0-56 from the Berg balance scale. A score of 56 means that the patient is independent and has no risk of falling. The closer the patient scores to "0 points", the higher the risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yu F, Evans LK, Sullivan-Marx EM. Functional outcomes for older adults with cognitive impairment in a comprehensive outpatient rehabilitation facility. J Am Geriatr Soc. 2005 Sep;53(9):1599-606. doi: 10.1111/j.1532-5415.2005.53453.x. PMID 16137294
- [Result] Sherrington C, Lord SR, Finch CF. Physical activity interventions to prevent falls among older people: update of the evidence. J Sci Med Sport. 2004 Apr;7(1 Suppl):43-51. doi: 10.1016/s1440-2440(04)80277-9. PMID 15214601
- [Result] Ghandali E, Moghadam ST, Hadian MR, Olyaei G, Jalaie S, Sajjadi E. The effect of Tai Chi exercises on postural stability and control in older patients with knee osteoarthritis. J Bodyw Mov Ther. 2017 Jul;21(3):594-598. doi: 10.1016/j.jbmt.2016.09.001. Epub 2016 Sep 10. PMID 28750970
- [Result] Xiong X, Wang P, Li S, Zhang Y, Li X. Effect of Baduanjin exercise for hypertension: a systematic review and meta-analysis of randomized controlled trials. Maturitas. 2015 Apr;80(4):370-8. doi: 10.1016/j.maturitas.2015.01.002. Epub 2015 Jan 9. PMID 25636242
- [Result] Zou L, Wang C, Chen X, Wang H. Baduanjin Exercise for Stroke Rehabilitation: A Systematic Review with Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2018 Mar 27;15(4):600. doi: 10.3390/ijerph15040600. PMID 29584623
- [Derived] Yildirim A, Hosbay Z, Ucgun H. The effect of Baduanjin exercise training on balance and fall risk in elderly individuals: A randomized controlled trial. Medicine (Baltimore). 2025 May 2;104(18):e42360. doi: 10.1097/MD.0000000000042360. PMID 40324224